CLINICAL TRIAL: NCT04798300
Title: Wear of Enamel Antagonist to Two Different Types of Monolithic Zirconia: A Randomized Clinical Trial
Brief Title: Wear of Enamel Antagonist to Two Different Types of Monolithic Zirconia Monolithic Zirconia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Ismail Mohamed Hussein, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 171020
Record Dates: First submitted 2021-01-28; First posted 2021-03-15 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Wear, Occlusal
MeSH Terms: conditions — Tooth Attrition

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tested material (Other): Newly Introduced Gradient Monolithic Zirconia (Intervention)
  Interventions: Procedure: Newly Introduced Gradient Monolithic Zirconia
- comparator material (Active Comparator): Full Strength Monolithic Zirconia (Comparator)
  Interventions: Procedure: Full Strength Monolithic Zirconia

INTERVENTIONS:
Procedure: Newly Introduced Gradient Monolithic Zirconia — Fabrication of full-coverage crowns over posterior teeth using Newly Introduced Gradient Monolithic Zirconia to measure wear
  Arms: tested material
Procedure: Full Strength Monolithic Zirconia — Fabrication of full-coverage crowns over posterior teeth using Full Strength Monolithic Zirconia to measure wear
  Arms: comparator material

SUMMARY:
The aim of the present study is to evaluate the wear of enamel opposed by Newly Introduced Gradient Monolithic Zirconia compared to that of enamel opposed by Full Strength Monolithic Zirconia

DETAILED DESCRIPTION:
The aim of the present study is to evaluate the wear of enamel opposed by Newly Introduced Gradient Monolithic Zirconia compared to that of enamel opposed by Full Strength Monolithic Zirconia Teeth preparation and impressions, placement and permanent cementation of the final restoration using resin cement, and optical scanning of both the restoration and the opposing tooth. Follow up postoperatively after six and twelve months, and optical scanning of both the restoration and the opposing tooth.

ELIGIBILITY:
Inclusion Criteria:

-

All subjects are required to be:

1. From 18-50 years old, be able to read and sign the informed consent document.
2. Have no active periodontal or pulpal diseases, have teeth with good restorations.
3. Psychologically and physically able to withstand conventional dental procedures.
4. Patients planned for a single coverage restoration in the posterior area.
5. Patients with a natural (not crowned) opposing antagonist.
6. Able to return for follow-up examinations and evaluation.

Exclusion Criteria:

* Patient less than 18 or more than 50 years 2. Patients with severe clenching or bruxing habits. 3. Patient with active resistant periodontal diseases 4. Patients with poor oral hygiene and uncooperative patients 5. Pregnant women 6. Patients in the growth stage with partially erupted teeth 7. Psychiatric problems or unrealistic expectations 8. Lack of opposing dentition at the area of interest. 9. Presence of dental prosthesis in the opposing arch at the area of interest.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Enamel wear of teeth opposing the restorations to be tested opposing to tested restorations | one year
  measured by Geomagic professional software

SECONDARY OUTCOMES:
Wear of restorations to tested opposed to natural teeth | one year
  measured by Geomagic professional software

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR